CLINICAL TRIAL: NCT05927129
Title: Research on the Biological Mechanism of the Efficacy of Psychotherapy for Depression Based on the Near-Infrared Functional Imaging System (fNIRS)
Brief Title: Research on the Biological Mechanism of the Efficacy of Psychotherapy for Depression Based on the fNIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-KY1-001-070
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Depressive Disorder
Keywords: Functional Near-Infrared Spectroscopy; fNIRS; depression; Biological Mechanism; Psychotherapy
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Antidepressive Agents; adenylate isopentenyltransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- medication therapy group (Active Comparator): Patients randomized to the medication therapy group will receive standardized treatment with antidepressant medications according to clinical guidelines.
  Interventions: Drug: Antidepressant
- Interpersonal Psychotherapy group (Active Comparator): The participants will receive standardized IPT treatment for 12 weeks. IPT therapists have received training from IPT workshops in both China and the United States and obtained the corresponding certifications. IPT therapists focus on the interpersonal domains associated with the onset and maintenance of depression. They guide clients in identifying the connections between their emotional changes and interpersonal difficulties, exploring problems, actively seeking potential interpersonal support and assistance, improving interpersonal skills, helping clients alleviate symptoms, enhance their quality of life, and adapt better to society.
  Interventions: Other: Psychotherapy IPT
- combination of medication therapy and Interpersonal Psychotherapy group (Experimental): Patients randomized to this group will receive standardized treatment with antidepressant medications according to clinical guidelines. The participants will also receive standardized IPT treatment for 12 weeks. IPT therapists have received training from IPT workshops in both China and the United States and obtained the corresponding certifications. IPT therapists focus on the interpersonal domains associated with the onset and maintenance of depression. They guide clients in identifying the connections between their emotional changes and interpersonal difficulties, exploring problems, actively seeking potential interpersonal support and assistance, improving interpersonal skills, helping clients alleviate symptoms, enhance their quality of life, and adapt better to society.
  Interventions: Other: The combination of antidepressant and IPT

INTERVENTIONS:
Drug: Antidepressant — Patients will receive standardized treatment with antidepressant, and their treatment efficacy will be assessed by a blinded psychological assessor using validated rating scales. The assessment will be conducted monthly, and evaluations will be tracked for a period of three months.
  Arms: medication therapy group
Other: Psychotherapy IPT — The participants will receive standardized IPT treatment for 12 weeks. Patients will receive standardized treatment, and their treatment efficacy will be assessed by a blinded psychological assessor using validated rating scales. The assessment will be conducted monthly, and evaluations will be tracked for a period of three months.
  Arms: Interpersonal Psychotherapy group
Other: The combination of antidepressant and IPT — The participants will receive standardized IPT treatment for 12 weeks. Also，long-term antidepressant will be administered in accordance with clinical guidelines. Patients will receive standardized treatment, and their treatment efficacy will be assessed by a blinded psychological assessor using validated rating scales. The assessment will be conducted monthly, and evaluations will be tracked for a period of three months.
  Arms: combination of medication therapy and Interpersonal Psychotherapy group

SUMMARY:
In this project, the investigators will implement medication therapy, psychotherapy, and a combination of medication therapy with psychotherapy, specifically utilizing IPT, in patients with depression. Simultaneously, the investigators will conduct comprehensive fNIRS assessments on all patients to evaluate changes in their brain function and determine the level of effectiveness of psychotherapy. The investigators will also employ standardized psychological assessments to evaluate patients, allowing for a comparison of the effectiveness of fNIRS assessments and providing clarity on the efficacy of psychotherapy in patients with depression, as the investigatorsll as the differential efficacy of different treatment approaches, and establishing the biological markers of psychotherapy. Additionally, the investigators will collect blood samples, cranial magnetic resonance images, and electroencephalograms from patients before and after treatment, which will contribute to further exploration of treatment mechanisms in the future.

DETAILED DESCRIPTION:
This study utilizes the Near-Infrared Functional Imaging System (fNIRS) as a biological marker for psychotherapy. The investigators propose the following scientific hypothesis: In patients with depression, levels of oxygenated hemoglobin and deoxygenated hemoglobin in different brain regions may fluctuate at different stages of the disease progression and treatment, along with changes in the activation levels of different brain regions. Neuroimaging studies on the neurobiological mechanisms of depression suggest a reduction in gray matter volume in emotion processing areas such as the limbic system, hippocampus, anterior cingulate cortex, dorsolateral prefrontal cortex, and basal ganglia. Previous neuroimaging studies have found that successful cognitive-behavioral therapy (CBT) accompanied changes in gray matter volume in the brain, as observed through fMRI. Interpersonal Psychotherapy (IPT), which is a component of the third wave of CBT, is expected to exhibit more significant expression in cognitive task-based fNIRS during IPT treatment for depression.

In this project, the investigators will implement medication therapy, psychotherapy, and a combination of medication therapy with psychotherapy, specifically utilizing IPT, in patients with depression. Simultaneously, the investigators will conduct comprehensive fNIRS assessments on all patients to evaluate changes in their brain function and determine the level of effectiveness of psychotherapy. The investigators will also employ standardized psychological assessments to evaluate patients, allowing for a comparison of the effectiveness of fNIRS assessments and providing clarity on the efficacy of psychotherapy in patients with depression, as the investigatorsll as the differential efficacy of different treatment approaches, and establishing the biological markers of psychotherapy. Additionally, the investigators will collect blood samples, cranial magnetic resonance images, and electroencephalograms from patients before and after treatment, which will contribute to further exploration of treatment mechanisms in the future.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for depression according to the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition).
* Have at least a junior high school education or higher.
* Age between 16 and 50 years old.
* Grew up in a Chinese-speaking environment and are proficient in Mandarin Chinese for effective communication.

Exclusion Criteria:

* Physical illnesses that significantly impact communication and mobility.
* Co-occurring psychiatric disorders other than depression.
* History of substance dependence or substance addiction.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in fNIRS (functional Near-Infrared Spectroscopy) after treatment. | Baseline, 4-weeks, 8-weeks,12-weeks.
  The instrument used in this study is a 52-channel Near-Infrared Spectroscopy (fNIRS) brain imaging system. It indirectly calculates the relative changes in levels of oxygenated and deoxygenated hemoglobin in different brain regions by detecting two different wavelengths of near-infrared light (695 nanometers and 830 nanometers). These changes reflect alterations in brain function. The instrument primarily utilizes 17 optical emitters and 16 optical detectors to acquire data. The emitters and detectors are positioned 3.0 centimeters apart, and the measurement area between the probes is defined as a channel. The NIRS probes are arranged in a 3×11 matrix, forming 52 measurement channels. Following the international 10-20 system, the lowest channel is aligned with the Fp1-Fp2 line. The probe coverage of this instrument allows for the measurement of relative changes in oxygenated and deoxygenated hemoglobin signals in bilateral frontal and temporal cortical regions.
Change in remission rate of Hamilton Depression Scale (24-items) (HAM-D24) score after treatment. | Baseline, 4-weeks, 8-weeks,12-weeks.
  The Hamilton Depression Scale (24-items) (HAM-D24), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4.
  Remission is defined as HAM-D24 ≤8.

SECONDARY OUTCOMES:
Change in remission rate of Patient Health Questionnaire-9 (PHQ-9) score after treatment. | Baseline, 4-weeks, 8-weeks,12-weeks.
  The Patient Health Questionnaire-9 (PHQ-9) is a screening tool used to assess symptoms of depression. It consists of nine questions that are designed to measure the severity of depressive symptoms experienced by an individual. Each question corresponds to one of the nine criteria for major depressive disorder as outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Each question is scored on a scale from 0 to 3, with higher scores indicating greater severity of symptoms. The total score ranges from 0 to 27, with higher scores indicating a higher likelihood of clinical depression. The PHQ-9 is widely used in both clinical and research settings to assess the presence and severity of depressive symptoms, monitor treatment progress, and aid in the diagnosis of depression.
Change in remission rate of the Beck Depression Inventory (BDI) score after treatment. | Baseline, 4-weeks, 8-weeks,12-weeks.
  The Beck Depression Inventory (BDI) is a widely used self-assessment tool for screening depression. Developed by American psychologist Aaron T. Beck in 1961, it aims to measure the severity of depressive symptoms experienced by an individual.
  The BDI consists of 21 items, each describing different aspects of depressive symptoms such as mood, loss of interest in activities, self-evaluation, changes in weight, sleep quality, and more. Individuals are required to rate their experiences based on a four-point scale ranging from 0 to 3, reflecting the intensity of each symptom.
  The total score on the BDI can range from 0 to 63, with higher scores indicating more severe depressive symptoms. The questionnaire is designed to assess the presence and severity of depression, monitor treatment progress, and aid in the diagnosis of depression.
Change in remission rate of the Beck Scale for Suicidal Ideation (SSI) score after treatment. | Baseline, 4-weeks, 8-weeks,12-weeks.
  The Beck Scale for Suicidal Ideation (SSI) is a self-report questionnaire designed to assess the presence and severity of suicidal thoughts and ideation. It was developed by Aaron T. Beck, a renowned psychologist, to aid in the evaluation of suicidal risk.
  The SSI consists of 19 items that explore different dimensions of suicidal ideation, including the intensity, frequency, duration, and specificity of suicidal thoughts. The questionnaire assesses both passive (e.g., "I wish I were dead") and active (e.g., "I have a plan to kill myself") suicidal ideation.
  Each item is rated on a scale from 0 to 2, with higher scores indicating a greater severity of suicidal ideation. The total score on the SSI can range from 0 to 38, providing an overall assessment of the individual's suicidal thoughts.

OTHER OUTCOMES:
Change in the score of THINC-it. | Baseline, 4-weeks, 8-weeks,12-weeks.
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it includes a series of brief tests that evaluate several cognitive domains, including attention, working memory, executive function, and processing speed. The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in neuroimaging using functional magnetic resonance | Baseline, 12-weeks.
  Scanning functional magnetic resonance. Functional magnetic resonance imaging (fMRI) is a neuroimaging technique that is used to measure changes in brain activity by detecting changes in blood flow. In the context of depression, fMRI has been used to study changes in brain function that may be associated with the condition. Research using fMRI in depression has shown that there are alterations in the activity of certain brain regions in people with the condition. Specifically, fMRI studies have identified changes in the activity of the prefrontal cortex, the amygdala, and the hippocampus in people with major depression. Overall, fMRI has provided valuable insights into the neural mechanisms underlying major depression, and may help to inform the development of new treatments for the condition.
Change in electroencephalogram | Baseline, 12-weeks.
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with depression and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of depression. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition.
Change of blood factor levels | Baseline, 8weeks, 12-weeks.
  Factors carried by peripheral blood and exosomes. The factors include brain-derived neurotrophic fact, Reelin and other reported factors related to depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Zhejiang, Hangzhou, China